CLINICAL TRIAL: NCT02489916
Title: Donafenib Monotherapy for Previously Treated Metastatic Colorectal Cancer: Multicentre, Open-label,Phase 1B Safety Study
Brief Title: Donafenib Monotherapy for Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGDC1B
Record Dates: First submitted 2014-09-28; First posted 2015-07-03 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2014-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; CM4307; Previously treated metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CM4307 (Experimental): CM4307 300mg bid，until disease progression,death, unacceptable toxic eff ects, withdrawal of consent by the patient, or decision by the treating physician that discontinuation would be in the patient's best interest
  Interventions: Drug: CM4307

INTERVENTIONS:
Drug: CM4307 — CM4307 300mg bid, each 4 week cycle
  Other Names: Donafenib

SUMMARY:
The investigators do the clinical trial (patients with metastatic colorectal cancer treated with donafenib after failure of standard therapy) to assess safety and efficacy of donafenib in patients with metastatic colorectal cancer, progressing after all approved standard therapies.

DETAILED DESCRIPTION:
The study is a multicentre, phase 1B study recruiting 47 patients in 6 sites. Patients were eligible to participate when they have histological or cytological documentation of adenocarcinoma of the colon or rectum. They must have received locally and currently approved standard therapies and to have disease progression during or within 3 months after the last administration of the last standard therapy or to have stopped standard therapy because of unacceptable toxic effects. The available standard therapies have to include as many of the following as were licensed: a fluoropyrimidine,oxaliplatin, irinotecan, and bevacizumab;and cetuximab or panitumumab for patients who had KRAS wild-type tumours.

Patients have to be aged 18 years or older and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; life expectancy of at least 3 months;and adequate bone-marrow, liver, and renal function at the start of the trial. Patients could not participate if they had previously received sorafenib or had uncontrolled medical disorders.

All patients receive best supportive care, excluding other investigational antitumour agents or antineoplastic chemotherapy, hormonal therapy, or immunotherapy. Patients receive oral donafenib 300mg (CM4307) of each 4 week cycle until disease progression,death, unacceptable toxic effects, withdrawal of consent by the patient, or decision by the treating physician that discontinuation would be in the patient's best interest.The primary endpoint is safety.The second endpoint is progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological documentation of adenocarcinoma of the colon or rectum;
* Have received locally and currently approved standard therapies and to have disease progression during or within 3 months after the last administration of the last standard therapy or to have stopped standard therapy because of unacceptable toxic effects.
* Standard therapies including as many of the following as were licensed: a fluoropyrimidine,oxaliplatin, irinotecan, and bevacizumab;and cetuximab or panitumumab for patients who had KRAS wild-type tumours;
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Life expectancy of at least 3 months;
* Have adequate bone-marrow, liver, and renal function at the start of the trial.
* Prothrombin time international normalized ratio≤2；or prothrombin time≤16 seconds;or activated partial thromboplastin time(APTT) ≤43 seconds;or TT≤21 seconds.

Exclusion Criteria:

* Patients have prior treatment with sorafenib;
* Patients have Central nervous system(CNS) involvement;
* patients have uncontrolled medical disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 54 weeks

SECONDARY OUTCOMES:
Progression Free Survival | 54 weeks

OTHER OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Feng Bi, Doctor, Principal Investigator — West China Hospital,SCU
Locations (1):
- West China Hospital,SCU, Chengdu, Sichuan, China